CLINICAL TRIAL: NCT06295224
Title: Retrospective Evaluation of Postoperative Analgesia Efficacy of the Anterior Iliac Block in Anterior Iliac Crest Bone Graft Harvesting: Preliminary Study
Brief Title: Retrospective Evaluation of Effect of Anterior Iliac Block
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hadi Ufuk Yörükoğlu, principal investigator, Kocaeli University
Other Study IDs: GOKAEK-2024/02.19
Record Dates: First submitted 2024-02-19; First posted 2024-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Regional Anesthesia
Keywords: Anterior Iliac Block; Anterior Iliac Crest Bone Harvesting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anterior Iliac Block: Patients who were performed anterior iliac block with ultrasound guidance with 10-20 mL 0.25% bupivacaine.

SUMMARY:
In this study, the investigators aimed to evaluate the effect of ultrasound-guided anterior iliac block which was performed preoperatively. Anterior iliac bone harvesting is associated with severe postoperative pain. As several fascial plane blocks were defined to provide analgesia, their effects are debatable and requires high volumes of local anesthetic considering the regional anesthesia technique used for the main surgical procedure.

DETAILED DESCRIPTION:
Autologous bone grafting is the method called the gold standard in the reconstruction of bone defects and nonunions. Anterior iliac crest is most frequently preferred as the source of autologous bone graft. However, severe pain after anterior iliac crest graft harvesting increases morbidity. Various regional anesthesia techniques have been defined for the purpose of postoperative analgesia. The mechanism of fascial plane blocks, one of these techniques, has not been fully elucidated and drug distribution varies from person to person. Postoperative analgesia of the iliac crest donor site can be achieved by i infiltration of local anesthetics or morphine. Single injection or continuous infusions of local anesthetic have proven effective in adults.

In this study; the investigators aimed to retrospectively scan the records of patients who received anterior iliac bone graft in our clinic and determine the postoperative analgesia effectiveness of anterior iliac block. The data obtained after the research will make a significant contribution to the literature in the postoperative analgesia management of patients who are planned to receive anterior iliac bone graft.

ELIGIBILITY:
Inclusion Criteria:

* ASA-1, ASA-2 and ASA-3 patients
* Female/male

Exclusion Criteria:

* Anticoagulant drug use
* Known allergy to the medications to be used
* Infection in the area where the needle will be inserted
* Missing data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent anterior iliac graft harvesting and were performed anterior iliac block at Kocaeli University Faculty of Medicine between January 2021 and December 2023 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | postoperative 1st hour, 6th hour, 12th hour and 24th hour
  Morphine consumption with patient controlled analgesia device

SECONDARY OUTCOMES:
NRS score | postoperative 1st hour, 6th hour, 12th hour and 24th hour
  NRS score at rest

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Ufuk Yörükoğlu, Principal Investigator — Kocaeli University, Department of Anesthesiology and Reanimation
Locations (1):
- Kocaeli Universty, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan SJ, Jeray KJ, Saliman LH, Miller HJ, Williams AE, Tanner SL, Smith WR, Broderick JS. Continuous infusion of local anesthetic at iliac crest bone-graft sites for postoperative pain relief. A randomized, double-blind study. J Bone Joint Surg Am. 2006 Dec;88(12):2606-12. doi: 10.2106/JBJS.E.00984. PMID 17142410
- [Background] Black ND, Malhas L, Jin R, Bhatia A, Chan VWS, Chin KJ. The analgesic efficacy of the transversalis fascia plane block in iliac crest bone graft harvesting: a randomized controlled trial. Korean J Anesthesiol. 2019 Aug;72(4):336-343. doi: 10.4097/kja.d.18.00352. Epub 2019 Mar 19. PMID 30886131
- [Background] Shin SR, Tornetta P 3rd. Donor Site Morbidity After Anterior Iliac Bone Graft Harvesting. J Orthop Trauma. 2016 Jun;30(6):340-3. doi: 10.1097/BOT.0000000000000551. PMID 27218470
- [Background] Sondekoppam RV, Ip V, Johnston DF, Uppal V, Johnson M, Ganapathy S, Tsui BCH. Ultrasound-guided lateral-medial transmuscular quadratus lumborum block for analgesia following anterior iliac crest bone graft harvesting: a clinical and anatomical study. Can J Anaesth. 2018 Feb;65(2):178-187. doi: 10.1007/s12630-017-1021-y. Epub 2017 Nov 21. PMID 29164530
- [Background] Gundes H, Kilickan L, Gurkan Y, Sarlak A, Toker K. Short- and long-term effects of regional application of morphine and bupivacaine on the iliac crest donor site. Acta Orthop Belg. 2000 Oct;66(4):341-4. PMID 11103484
- [Background] Chin KJ, McDonnell JG, Carvalho B, Sharkey A, Pawa A, Gadsden J. Essentials of Our Current Understanding: Abdominal Wall Blocks. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):133-183. doi: 10.1097/AAP.0000000000000545. PMID 28085788
- [Background] Ouaki J, Dadure C, Bringuier S, Raux O, Rochette A, Captier G, Capdevila X. Continuous infusion of ropivacaine: an optimal postoperative analgesia regimen for iliac crest bone graft in children. Paediatr Anaesth. 2009 Sep;19(9):887-91. doi: 10.1111/j.1460-9592.2009.03095.x. PMID 19691695
- [Derived] Yorukoglu HU, Cesur S, Izgin Avci I, GoK A, Aksu C, Selek O, Kus A. Retrospective evaluation of postoperative analgesia efficacy of a new technique in anterior iliac crest bone graft harvesting: anterior iliac block. BMC Anesthesiol. 2024 Nov 29;24(1):443. doi: 10.1186/s12871-024-02829-7. PMID 39609729